CLINICAL TRIAL: NCT03458052
Title: Knowledge, Professional Experience and Attitude Toward Organ Donation Among Health Care Professionals in Argentina: the DonAR Survey
Brief Title: Organ Donation Survey Among Health Care Professionals in Argentina
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: 3493
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Brain Death; Lung Transplantation; Respiration, Artificial; Tissue and Organ Procurement
Keywords: Intensive and critical care; Organ donation; Knowledge
MeSH Terms: conditions — Brain Death; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to gather information about knowledge, professional experience and attitude toward organ donation among health care professionals involved in the care of potential donors about the procurement process and potential lung donor management nationwide.

DETAILED DESCRIPTION:
The shortage of cadaveric organ donors for transplantation is a global problem. This fact prolongs the time on the waiting list and, therefore, the mortality, which rise to 21.15% in Argentina compared to a world average of 16%. Many reasons can explain the low procurement rate. It has been stated that the conventional ventilatory management for potential lung donors is suboptimal for lung preservation before harvest.

In Argentina there is limited research regarding the attitude toward organ donation among health care professionals, knowledge of the federal organ procurement program and professional experience in diagnosing brain death and lung donor management. Knowing the Argentinian current situation will make it possible to detect possible organ shortages causes, evaluate strategies to increase the national procurement rate and to instruct the health team that assists neurocritical patients who die of brain death. So we propose the following research.

The aim of this study is to gather information about knowledge, professional experience and attitude among health care professionals involved in the care of potential donors toward organ donation, procurement process and potential lung donor management nationwide.

A online questionnaire was designed and distributed among health care professionals register to different scientific societies related to the care of neurocritical patients between febrary 16th and september 1st. The questionnaire consisting of 37 ítems: 6 items measuring attitudes, 6 items measuring knowledge, 16 items investigating professional experience and 9 ítems assessing demographics.

ELIGIBILITY:
Inclusion Criteria:

* health care professionals
* register to the Sociedad Argentina de Terapia Intensiva (SATI)
* related to the care of neurocritical patients
* between febrary 16th and september 1st.

Exclusion Criteria:

* unrelated to the care of neurocritical patients

Ages: 23 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heath Care Professionals working in Adult and Pediatric Critical Care Units and Emergency Department from Argentinian Public and Private Hospitals, registrated in the Sociedad Argentina de Terapia Intensiva
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Attitude Toward Organ Donation | 6 months
  investigated attitudes regarding organ donation among health care professional: is an organ donor:1, isn´t an organ donor:2, he/she haven´t been decided: 2
Organ Donor Registry | 6 months
  investigated whether the health care professional is a registered organ donor: Yes:1, No:0.
Last will manifest | 6 months
  investigated whether the health care professional´s spouse and / or family knows he/she organ donor attitude towards organ donation: Yes:1, No:0.
Reasons to donate | 6 months
  investigated reasons why the health care professional´ would donate their organs: To save the life of another person: 1, Because after death the body does not need anything: 2, To create awareness in the donation: 3, For religious reasons: 4, Others: 5
Reasons not to donate | 6 months
  investigated reasons why the health care professional´ would not donate their organs or haven´t decided: for religious aspects: 1, for the improper organs use: 2, to maintain my body integrity: 3, for fear of the removal of organs before my death: 4, for fear that they do not give me the attention Medical needed to save my life: 5, Others: 6
Level of knowledge | 6 months
  investigated how the health care professional would classify the level of knowledge regarding organ donation: Not at all informed: 1, Little informed: 2, Suitably informed: 3
Degree formation | 6 months
  investigated whether the health care professional received organ donation information during their degree formation: Yes:1, No:0.
Post degree formation | 6 months
  investigated whether the health care professional attended to courses on procurement or organ donation after their degree formation: Yes:1, No:0.
Brain death definition | 6 months
  investigated when health care professional consider a neurocritical patient as a potential organ donor: When the patient is in a coma: 1, When brain inactivity is corroborated with technical or instrumental means in a patient with irreversible absence of brain response with loss of consciousness, absence of spontaneous breathing, absence of cephalic reflexes and observation of fixed pupils: 2, When the patient is in a vegetative state: 3, When cardiorespiratory arrest occurs in the patient with irreversible absence of brain response with loss of consciousness, absence of spontaneous breathing, absence of cephalic reflexes and fixation of fixed pupils: 4, Other: 5
Lung organ donor criteria | 6 months
  investigated whether the health care professional know the criteria the organ donor must meet to be considered an optimal lung donor. PaO2 / FiO2> 300 with FiO2 1 and PEEP 10cmH2O, without evidence of aspiration / sepsis, absence of microorganism in sputum / BAL, absence of purulent secretions in tube: 1, X-ray with minimal infiltrates, no evidence of aspiration / sepsis, no history of cardiopulmonary surgery, absence of microorganism in sputum / BAL, absence of secretions: 2, clean chest X-ray, PaO2 / FiO2> 300 with FiO2 1 and PEEP 5cmH2O, absence of thoracic trauma, without evidence of aspiration / sepsis, no history of cardiopulmonary surgery, absence of microorganism in sputum / BAL, absence of purulent secretions in tube: 3, d. Unilateral thoracic trauma, with no evidence of aspiration / sepsis, no history of cardiopulmonary surgery, absence of microorganism in sputum / BAL, absence of purulent secretions in tube: 4
Organ Donor Consent | 6 months
  investigated whether the health care professional knows where and how to express he/she consent for organ donation: Yes:1, No:0.
Potential lung donor management protocols | 6 months
  investigated whether the health care professional knows if the health care institution were he/she works have a potential lung donor management protocol.
Neurocritical patients care | 6 months
  investigated whether the health care professional had ever assist a neurocritical patients during this professional career.
Call to the federal organ procurement organism to report a patients with a GCS ≤ 7 | 6 months
  investigated whether the health care professional had ever call to the federal organ procurement organism (INCUCAI) to report a neurocritical patients with a GCS ≤ 7.
Apnea Test | 6 months
  investigated whether the health care professional had ever done an apnea test during this professional career.
Type of apnea test | 6 months
  investigated which type of apnea test the health care professional had done: the conventional apnea test consisting in preoxygenation and disconnection form the ventilator; or one of the alternative apnea test: by artificial increase of Co2; with CPAP or by controlled hypoventilation.
Call to the federal organ procurement organism to report a possible brain death patient: | 6 months
  investigated whether the health care professional had ever call to the federal organ procurement organism (INCUCAI) to report a possible brain death patient.
Potential organ donor patients care | 6 months
  investigated whether the health care professional had ever participated in the procurement process and maintenance (management) of a potential organ donor patient during this professional career.
Change in ventilator parameters | 6 months
  investigated whether the health care professional make a change in the ventilator parameters after the brain dead diagnosis.
Change in the fraction inspired oxygen | 6 months
  investigated whether the health care professional change the fraction inspired oxygen to 100% after the brain dead diagnosis, or reduced it if the potential lung donor have a PaO2/FiO2 > 300.
Ventilator parameters | 6 months
  investigated which tidal volume (Vt) and positive end expiratory pressure (PEEP) does the health care professional use to ventilate a potential lung donor patient among different options: Vt 10-12 mL/kg, PEEP 5 cmH20:1, Vt 10-12 mL/kg, PEEP 8-10 cmH20:2, Vt 8-10 mL/kg, PEEP 5 cmH20:3, Vt 8-10 mL/kg, PEEP 8-10 cmH20:4, Vt 6-8 mL/kg, PEEP 5 cmH20:5, Vt 6-8 mL/kg, PEEP 8-10cmH20:6, Other:7
Strategies to improve oxygenation | 6 months
  investigated whether the health care professional use any strategy to improve oxygenation in case of low oxygenation and which type of strategies does it use: change positioning:1, pulmonary expansion techniques:2, endotracheal suctioning:3, Fiberoptic bronchoscopy:4, Recruitment maneuvers: 5, PEEP titulation:6, Others:7
Type of Recruitment maneuver | 6 months
  investigated the most commonly used type of recruitment maneuver in a potential PULMONARY donor: Sighs with increased Tidal Volume for several breaths: 1, CPAP of 40 cmH20 for 40 seconds: 2, CPAP of 30 cmH20 for 30 seconds: 3, Step increase of PEEP to 40 cmH20 and then stepwise decrease: 4, PC Mode CMV with inspiratory pressure of 25-30 cmH20 and PEEP 10-15 cmH20 for 2 hours for a single time: 5, PC-CMV mode with inspiratory pressure of 20 cmH20 and stepwise increase of PEEP to 20-30 cmH20: 6, PEEP of 18-20 cmH20 for 1 minute, then decrease PEEP and increase Tidal Volume for several breaths: 7, Other: 8.
Type of PEEP titulation | 6 months
  PEEP / FiO2 Table (ARDS Network): 1, PEEP / Compliance Protocol: 2, Determination of the lower inflection point per Pressure / Volume curve: 3, Increase of the PEEP for Plateau Pressure <28 cmH20 (Express Protocol): 4, Guided by esophageal manometry: 5, Guided by pulmonary ultrasound: 6, Guided by volumetric capnography: 7, Other: 8
Use of a closed-circuit for endotracheal suctioning | 6 months
  investigated whether the health care professional use a closed-circuit for endotracheal suctioning.
Measures to prevent ventilator-associated pneumonia | 6 months
  investigated whether the health care professional consider important to continue the care bundle to prevent ventilator-associated pneumonia such as: head elevation, tracheal cuff control, oral hygiene, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa R Ruiz, RT, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Result] Minambres E, Coll E, Duerto J, Suberviola B, Mons R, Cifrian JM, Ballesteros MA. Effect of an intensive lung donor-management protocol on lung transplantation outcomes. J Heart Lung Transplant. 2014 Feb;33(2):178-84. doi: 10.1016/j.healun.2013.10.034. Epub 2013 Oct 25. PMID 24365763
- [Result] Mascia L, Mastromauro I, Viberti S, Vincenzi M, Zanello M. Management to optimize organ procurement in brain dead donors. Minerva Anestesiol. 2009 Mar;75(3):125-33. Epub 2008 Jan 24. PMID 18636057
- [Result] Valapour M, Paulson K, Smith JM, Hertz MI, Skeans MA, Heubner BM, Edwards LB, Snyder JJ, Israni AK, Kasiske BL. OPTN/SRTR 2011 Annual Data Report: lung. Am J Transplant. 2013 Jan;13 Suppl 1:149-77. doi: 10.1111/ajt.12024. PMID 23237700
- [Result] Del Rio F, Escudero D, De La Calle B, Vidal FG, Paredes MV, Nunez JR. [Evaluation and maintenance of the lung donor]. Med Intensiva. 2009 Jan-Feb;33(1):40-9. doi: 10.1016/s0210-5691(09)70304-3. Spanish. PMID 19232208
- [Result] Rosengard BR, Feng S, Alfrey EJ, Zaroff JG, Emond JC, Henry ML, Garrity ER, Roberts JP, Wynn JJ, Metzger RA, Freeman RB, Port FK, Merion RM, Love RB, Busuttil RW, Delmonico FL. Report of the Crystal City meeting to maximize the use of organs recovered from the cadaver donor. Am J Transplant. 2002 Sep;2(8):701-11. doi: 10.1034/j.1600-6143.2002.20804.x. No abstract available. PMID 12243491
- [Result] Mascia L, Bosma K, Pasero D, Galli T, Cortese G, Donadio P, Bosco R. Ventilatory and hemodynamic management of potential organ donors: an observational survey. Crit Care Med. 2006 Feb;34(2):321-7; quiz 328. doi: 10.1097/01.ccm.0000196828.87358.6e. PMID 16424709
- [Result] Mascia L, Pasero D, Slutsky AS, Arguis MJ, Berardino M, Grasso S, Munari M, Boifava S, Cornara G, Della Corte F, Vivaldi N, Malacarne P, Del Gaudio P, Livigni S, Zavala E, Filippini C, Martin EL, Donadio PP, Mastromauro I, Ranieri VM. Effect of a lung protective strategy for organ donors on eligibility and availability of lungs for transplantation: a randomized controlled trial. JAMA. 2010 Dec 15;304(23):2620-7. doi: 10.1001/jama.2010.1796. PMID 21156950
- [Result] Klesney-Tait JA, Eberlein M. Lung protective ventilation in donors: an ounce of prevention. Chest. 2014 Jul;146(1):4-6. doi: 10.1378/chest.14-0163. No abstract available. PMID 25010954
- [Result] McKeown DW, Bonser RS, Kellum JA. Management of the heartbeating brain-dead organ donor. Br J Anaesth. 2012 Jan;108 Suppl 1:i96-107. doi: 10.1093/bja/aer351. PMID 22194439
- [Result] Bansal R, Esan A, Hess D, Angel LF, Levine SM, George T, Raoof S. Mechanical ventilatory support in potential lung donor patients. Chest. 2014 Jul;146(1):220-227. doi: 10.1378/chest.12-2745. PMID 25010965
- [Result] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Result] Munshi L, Keshavjee S, Cypel M. Donor management and lung preservation for lung transplantation. Lancet Respir Med. 2013 Jun;1(4):318-28. doi: 10.1016/S2213-2600(12)70064-4. Epub 2013 Feb 20. PMID 24429157
- [Result] Lucangelo U, Del Sorbo L, Boffini M, Ranieri VM. Protective ventilation for lung transplantation. Curr Opin Anaesthesiol. 2012 Apr;25(2):170-4. doi: 10.1097/ACO.0b013e32834fdb54. PMID 22228421
- [Result] Al-Khafaji A, Murugan R, Kellum JA. What's new in organ donation: better care of the dead for the living. Intensive Care Med. 2013 Nov;39(11):2031-3. doi: 10.1007/s00134-013-3038-1. Epub 2013 Aug 3. No abstract available. PMID 23912380
- [Result] Angel LF, Levine DJ, Restrepo MI, Johnson S, Sako E, Carpenter A, Calhoon J, Cornell JE, Adams SG, Chisholm GB, Nespral J, Roberson A, Levine SM. Impact of a lung transplantation donor-management protocol on lung donation and recipient outcomes. Am J Respir Crit Care Med. 2006 Sep 15;174(6):710-6. doi: 10.1164/rccm.200603-432OC. Epub 2006 Jun 23. PMID 16799075
- [Result] Kirschbaum CE, Hudson S. Increasing organ yield through a lung management protocol. Prog Transplant. 2010 Mar;20(1):28-32. doi: 10.1177/152692481002000105. PMID 20397343
- [Result] Paries M, Boccheciampe N, Raux M, Riou B, Langeron O, Nicolas-Robin A. Benefit of a single recruitment maneuver after an apnea test for the diagnosis of brain death. Crit Care. 2012 Jul 3;16(4):R116. doi: 10.1186/cc11408. PMID 22759403
- [Result] Gabbay E, Williams TJ, Griffiths AP, Macfarlane LM, Kotsimbos TC, Esmore DS, Snell GI. Maximizing the utilization of donor organs offered for lung transplantation. Am J Respir Crit Care Med. 1999 Jul;160(1):265-71. doi: 10.1164/ajrccm.160.1.9811017. PMID 10390410
- [Result] Noiseux N, Nguyen BK, Marsolais P, Dupont J, Simard L, Houde I, Lallier M, Langevin S, Cantin B, Ferraro P. Pulmonary recruitment protocol for organ donors: a new strategy to improve the rate of lung utilization. Transplant Proc. 2009 Oct;41(8):3284-9. doi: 10.1016/j.transproceed.2009.08.041. PMID 19857731
- [Result] Hanna K, Seder CW, Weinberger JB, Sills PA, Hagan M, Janczyk RJ. Airway pressure release ventilation and successful lung donation. Arch Surg. 2011 Mar;146(3):325-8. doi: 10.1001/archsurg.2011.35. PMID 21422364
- [Result] Philpot SJ, Pilcher DV, Graham SM, Snell GI. Lung recruitment manoeuvres should be considered when assessing suitability for lung donation. Crit Care Resusc. 2012 Sep;14(3):244-5. No abstract available. PMID 22963221
- [Result] Parto S, Shafaghi S, Khoddami-Vishteh HR, Makki SM, Abbasidezfuli A, Daneshvar A, Sheikhy K, Faeghi J, Ghorbani F, Parsa T, Najafizadeh K. Efficacy of recruitment maneuver for improving the brain dead marginal lungs to ideal. Transplant Proc. 2013;45(10):3531-3. doi: 10.1016/j.transproceed.2013.09.001. PMID 24314951
- See also: Alejandro Da Lozzo. Historia del trasplante pulmonar en el mundo y en la Argentina. Rev Hosp Ital. B.Aires 2013;33(3):111-119. — https://www.hospitalitaliano.org.ar/multimedia/archivos/servicios_attachs/8936.pdf
- See also: Ruiz V. R., Da Lozzo A. G., Midley A. D. Optimización del Soporte Ventilatorio del Donante Pulmonar. Revisión Bibliográfica. RAMR 2017;2:174-179 — http://www.scielo.org.ar/pdf/ramer/v17n2/v17n2a14.pdf